CLINICAL TRIAL: NCT01459406
Title: Effects of FODMAPs (Fermentable Oligo-, Di-, and Mono-saccharides, And Polyols) on Small Bowel Water Content: an MRI Study
Brief Title: Effects of FODMAPs on Small Bowel Water Content: an MRI Study
Acronym: FODMAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: L/7/2011
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Gastrointestinal physiology; Gastrointestinal response to sugars; MRI; gastrointestinal; stomach; small bowel; colon; glucose; fructose; fructan; FODMAP
MeSH Terms: interventions — Glucose; Fructose; Fructans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glucose drink (Experimental): Serial MRI of the gastrointestinal tract upon 500 ml water drink containing 40g glucose
  Interventions: Dietary Supplement: Glucose
- Fructose drink (Experimental): Serial MRI of the gastrointestinal tract upon 500 ml water drink containing 40g fructose
  Interventions: Dietary Supplement: Fructose
- Fructan drink (Experimental): Serial MRI of the gastrointestinal tract upon 500 ml water drink containing 40g fructan
  Interventions: Dietary Supplement: Fructan
- Fructose and glucose drink (Experimental): Serial MRI of the gastrointestinal tract upon 500 ml water drink containing 40g fructose and 40 g glucose
  Interventions: Dietary Supplement: Fructose and glucose

INTERVENTIONS:
Dietary Supplement: Glucose — 500 ml water drink containing 40g glucose
  Arms: Glucose drink
Dietary Supplement: Fructose — 500 ml water drink containing 40g fructose
  Arms: Fructose drink
Dietary Supplement: Fructan — 500 ml water drink containing 40g fructan
  Arms: Fructan drink
Dietary Supplement: Fructose and glucose — 500 ml water drink containing 40g fructose and 40g glucose
  Arms: Fructose and glucose drink

SUMMARY:
Some carbohydrates, particularly fructose, the sugar found in fruit and bread may cause bloating, pain and erratic bowel habits (diarrhoea and constipation) particularly in patients suffering from the irritable bowel syndrome (IBS). This may be because they are not well absorbed in the small intestine and cause water to be trapped in the bowel causing distension. Studies have shown that reducing the amount of these sugars in the diet can relieve these symptoms. There is some evidence that combining fructose and glucose can reduce the symptoms caused by fructose but just why is unclear. In this study, the investigators will use a non invasive medical imaging technique called "magnetic resonance imaging" (or MRI) to look at the behaviour of drinks containing these sugars in the bowels of healthy human volunteers.

The investigators will give four different drinks: one beverage consisting of a very well absorbed sugar, glucose, another consisting of the less well absorbed sugar fructose, a third which is a mixture of glucose and fructose, and a fourth consisting of several fructose subunits joined together (called fructan). The investigators will take MRI images of the stomach and intestines at intervals for 5 hours and compare these with the feelings of distension and bloating in our volunteers. The results will act as control for subsequent studies in IBS patients and these may help design diets to reduce symptoms in IBS.

DETAILED DESCRIPTION:
Title: Effects of FODMAPs (Fermentable Oligo-, Di-, and Mono-saccharides, And Polyols) on small bowel water content: an MRI study

1. Background. FODMAPs consist of fructose, lactose, fructo- and galacto-oligosaccharides such as fructans and galactans, and polyols such as sorbitol and mannitol. These carbohydrates are poorly absorbed in the small intestine and have been shown to trigger symptoms of irritable bowel syndrome (IBS). Previous studies have shown that fructose malabsorption results in an increased osmotic load in the small bowel, which can have a laxative effect. Physical proof of this has only been obtained using an ileostomy model on patients. This study indicated increased small bowel water content (SBWC) but this has never been established in intact humans .). We have been using noninvasive magnetic resonance imaging (MRI) to provide novel insights on the fate of food materials within the gastro-intestinal tract (GIT) of humans for the last decade.
2. Aims (to include hypothesis to be tested) This study aims to investigate whether fructose alone will increase SBWC compared to an equivalent mass of glucose, and if adding glucose to fructose will reduce its effect on the SBWC. The study also aims to determine if fructans alter colonic transit.The main hypothesis is that fructose will increase small bowel water while fructans will mainly affect colonic transit..
3. Experimental protocol and methods. A single-centre, randomized, cross-over design study consisting of a screening visit and four test days, which will be approximately 1 week apart The subjects (18 healthy volunteers for main study plus 4 for pilot studies) will receive (according to a randomization schedule) each test day one out of four test products: 1) glucose (control) 2) fructose, 3) glucose with fructose and 4) fructans. On each test day, volunteers will have a baseline scan in a 1.5T scanner, consume one of the products instead of breakfast at 09:00 and will be imaged in the scanner at intervals for 5 hours using a range of MRI sequences.

All the tested ingredients are food grade, have a history of safe use at intended usage levels, and are regarded as safe.

Four test products will be evaluated:

1. 500 mL of glucose (40g of glucose dissolved in water with pure lime juice as flavorant)
2. 500 mL fructose (40g fructose dissolved in water with pure lime juice as flavorant)
3. 500 mL of glucose with fructose (40g glucose and 40g fructose dissolved in water with pure lime juice as flavorant, 40 or 80 gm)
4. 500 mL fructan (40g of 100% fructan (inulin) dissolved in water with pure lime juice as flavorant)

4. Measurable end points/statistical power of the study. Primary endpoint: small bowel water content area under the curve (AUC) -45 - 315 minutes. Secondary endpoint: gastric emptying T50, colonic volume as characterised by AUC -45 - 315 minutes of ascending colon, colonic motility, symptoms questionnaires, small bowel transit time, breath hydrogen concentrations and tryptase faecal content.

Previous work using mannitol and glucose indicates that mean (SD) SBWC at 40 minutes postprandial after ingesting 300ml glucose was 47 (SD 15) and using n=12 the investigators calculate the investigators can detect an increase of 20 ml in excess of this with 90% power which is very much less than the investigators are predicting. The investigators plan to use 18 to ensure the investigators can assess our secondary endpoints for which there is no data with which to perform a power calculation.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy: no medical conditions which might effect study measurements.
* No reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.
* Age ≥ 18 and ≤ 60 year at pre-study investigation.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2
* No reported participation in night shift work two days prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Strenuous exercise ≤ 10 hours per week.
* Gender: male or female
* Consumption of ≤ 21 alcoholic drinks in a typical week
* Currently not smoking
* Suitable for MRI scanning (e.g., absence of metal implants, infusion pumps and pacemakers) as assessed by the attached MRI safety questionnaire.

Exclusion Criteria:

* - use of medication which interferes with study measurements or bowel motility (as judged by the study physician).
* Antibiotics in the 3 weeks before pre-study examination
* Probiotics or during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
small bowel water content area under the curve | -45 min to 315 min
  Area Under the curve for small bowel water content, methods as Marciani, L., et al., Gastroenterology, 2010. 138(2): p. 469-U90. Hoad, C.L., et al.,. Physics in Medicine and Biology, 2007. 52(23): p. 6909-6922.

SECONDARY OUTCOMES:
gastric emptying T50 | -45 min to 315 min
  time to half empty the stomach
ascending colon volume | -45 min to 315 min
  AUC of the geometric volume of the ascending colon
ascending colon motility | -45 min to 315 min
  motility index of the ascending colon as determined from dynamic MRI scan
symptoms questionnaires | -45 min to 315 min
  bloating, nausea, gas belching and abdominal pain
bowel transit time | 24 hours
  first time to detect sweetcorn markers in the stool
fecal tryptase activity | 24 h
  activity of stool triptase in trypsin units of activity

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD FRCP, Principal Investigator — University of Nottingham
Locations (1):
- NDDC BRU and Sir Peter Mansfield Magnetic Resonance Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Ong DK, Mitchell SB, Barrett JS, Shepherd SJ, Irving PM, Biesiekierski JR, Smith S, Gibson PR, Muir JG. Manipulation of dietary short chain carbohydrates alters the pattern of gas production and genesis of symptoms in irritable bowel syndrome. J Gastroenterol Hepatol. 2010 Aug;25(8):1366-73. doi: 10.1111/j.1440-1746.2010.06370.x. PMID 20659225
- [Background] Marciani L, Cox EF, Hoad CL, Pritchard S, Totman JJ, Foley S, Mistry A, Evans S, Gowland PA, Spiller RC. Postprandial changes in small bowel water content in healthy subjects and patients with irritable bowel syndrome. Gastroenterology. 2010 Feb;138(2):469-77, 477.e1. doi: 10.1053/j.gastro.2009.10.055. Epub 2009 Nov 10. PMID 19909743
- [Background] Hoad CL, Marciani L, Foley S, Totman JJ, Wright J, Bush D, Cox EF, Campbell E, Spiller RC, Gowland PA. Non-invasive quantification of small bowel water content by MRI: a validation study. Phys Med Biol. 2007 Dec 7;52(23):6909-22. doi: 10.1088/0031-9155/52/23/009. Epub 2007 Nov 8. PMID 18029983
- [Background] Gibson PR, Barrett JS. The concept of small intestinal bacterial overgrowth in relation to functional gastrointestinal disorders. Nutrition. 2010 Nov-Dec;26(11-12):1038-43. doi: 10.1016/j.nut.2010.01.005. Epub 2010 Apr 24. PMID 20418060
- [Background] Shepherd SJ, Parker FC, Muir JG, Gibson PR. Dietary triggers of abdominal symptoms in patients with irritable bowel syndrome: randomized placebo-controlled evidence. Clin Gastroenterol Hepatol. 2008 Jul;6(7):765-71. doi: 10.1016/j.cgh.2008.02.058. Epub 2008 May 5. PMID 18456565
- [Background] Shepherd SJ, Gibson PR. Fructose malabsorption and symptoms of irritable bowel syndrome: guidelines for effective dietary management. J Am Diet Assoc. 2006 Oct;106(10):1631-9. doi: 10.1016/j.jada.2006.07.010. PMID 17000196
- [Background] Barrett JS, Gearry RB, Muir JG, Irving PM, Rose R, Rosella O, Haines ML, Shepherd SJ, Gibson PR. Dietary poorly absorbed, short-chain carbohydrates increase delivery of water and fermentable substrates to the proximal colon. Aliment Pharmacol Ther. 2010 Apr;31(8):874-82. doi: 10.1111/j.1365-2036.2010.04237.x. Epub 2010 Jan 22. PMID 20102355
- [Background] Khoshini R, Dai SC, Lezcano S, Pimentel M. A systematic review of diagnostic tests for small intestinal bacterial overgrowth. Dig Dis Sci. 2008 Jun;53(6):1443-54. doi: 10.1007/s10620-007-0065-1. PMID 17990113
- [Background] Rumessen JJ, Gudmand-Hoyer E. Fructans of chicory: intestinal transport and fermentation of different chain lengths and relation to fructose and sorbitol malabsorption. Am J Clin Nutr. 1998 Aug;68(2):357-64. doi: 10.1093/ajcn/68.2.357. PMID 9701194
- [Background] Bond JH Jr, Levitt MD, Prentiss R. Investigation of small bowel transit time in man utilizing pulmonary hydrogen (H2) measurements. J Lab Clin Med. 1975 Apr;85(4):546-55. PMID 1120927